CLINICAL TRIAL: NCT02111837
Title: Multicenter, Randomized, Double-blind, Parallel-group, Reference-controlled, Safety Pilot Study to Evaluate the Effects of Specific Lipid Fractions-enriched Infant Formulae in Infants Aged 0-4 Months
Brief Title: Effects of Specific Lipid Fractions-enriched Infant Formulae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 07.16.INF.B
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Infant Growth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard infant formula (Placebo Comparator): Standard infant formula fed ad libitum
  Interventions: Other: Standard infant formula
- Standard infant formula with PL1 (Experimental): Standard infant formula enriched with PL1 lipid fraction fed ad libitum
  Interventions: Other: Standard infant formula with PL1
- Standard infant formula with PL2 (Experimental): Standard infant formula enriched with PL2 lipid fraction fed ad libitum
  Interventions: Other: Standard infant formula with PL2

INTERVENTIONS:
Other: Standard infant formula
  Arms: Standard infant formula
Other: Standard infant formula with PL1
  Arms: Standard infant formula with PL1
Other: Standard infant formula with PL2
  Arms: Standard infant formula with PL2

SUMMARY:
This is a multicenter, randomized, double-blind, parallel-group, reference-controlled 4-month pilot safety study to evaluate the effects of specific lipid fractions-enriched infant formulae on growth of infants aged 0-4 months. The study will test the hypothesis that growth of infants fed the specific lipid fractions-enriched infant formulae will be noninferior to growth of infants fed standard infant formula.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn infant
* Infant is ≤14 days old on day of enrollment
* Gestational age ≥37 weeks (full term infants)
* Birth weight ≥2500 g and ≤4500 g
* Singleton birth
* Having obtained his/her parents'/legal representative's informed consent

Exclusion Criteria:

* Having any significant pre-natal and/or post-natal disease and/or congenital illness or malformation that may affect normal growth.
* Infant undergoing antibiotic therapy.
* Re-hospitalization for more than 2 days in the first 14 days of life.
* Parents not expected to comply with the protocol during the period of study participation.
* Infants currently participating in another trial

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 199 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Mean weight gain (g/day) | Enrollment to age 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Claude Billeaud, MD, Principal Investigator — Hôpital des enfants, CHU Pellegrin, Bordeaux, France
Locations (4):
- France (3):
  - CHU de Caen, Caen, Cedex 9
  - Hôpital Bretonneau - UPM, Tours, Cedex 9
  - Groupe Hospitalier Pellegrin, Bordeaux
- Istituto di Ostetricia e Ginecologia Neonatalogia, Palermo, Italy